CLINICAL TRIAL: NCT02618109
Title: Identification of New Immune Factors Specific of Relapse in Childhood B Lineage Acute Lymphoblastic Leukemia
Acronym: LABMI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-A00621-48
Record Dates: First submitted 2015-04-15; First posted 2015-12-01 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: B Acute Lymphoblastic Leukemia; Leukemia Relapse
Keywords: B acute lymphoblastic leukemia; leukemia relapse; pediatric onco-hematology
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relapse Group (Other): * Collection of blood samples will be done in newly diagnosed relapse of B-ALL children at the time of relapse diagnosis.
  * Children aged from 1 to 18 years at the time of first B-ALL relapse diagnosis.
  Interventions: Biological: Collection of blood samples
- Control Group (Other): * Collection of blood samples will be done at the same stage of treatment as the relapse group has been collected.
  * Children aged from 1 to 18 years enrolled into FRALLE (protocol of treatment) or EORTC (European Organisation for Research and Treatment of Cancer) treatment protocols, treated for B-ALL and who are in complete molecular remission.
  * These control patients will be recruited at the same time from the beginning of B-ALL treatment as paired-relapsed control patients.
  Interventions: Biological: Collection of blood samples

INTERVENTIONS:
Biological: Collection of blood samples — Collection of blood samples

SUMMARY:
B-acute lymphoblastic leukaemia (ALL) is the most common childhood malignancy. Despite enhancement of childhood B-ALL outcome, relapses remain difficult to treat. Several studies in adult acute myeloid leukaemia have shown that proliferation of immunosuppressive cells -particularly T regulatory (Treg) cells and deficient natural killer (NK) cells- was associated with poor response to chemotherapy. However, few studies have been done on childhood ALL and none on relapse of B-ALL. Moreover, a newly described immunosuppressive B cells subset (Breg cells) seems to have a role in oncogenesis in mice model, but its significance has never been evaluated in human cancers. The purpose of this study is to prospectively evaluate the immune status of children newly diagnosed with first relapse of B-cell ALL, and to compare results with those of children treated for B-ALL in complete remission. Classic lymphocytic phenotype, proportions of immunosuppressive cells (Treg cells, deficient NK cells, Cytotoxic T-lymphocyte-associated protein 4 and/or Programmed T cell death 1) and thymopoiesis will be evaluated. The investigators assume that increase of immunosuppressive cells proportions could be associated with B-ALL relapse.

ELIGIBILITY:
1. Inclusion Criteria for relapse Group :

   * Children aged from 1 to 18 years at the time of first B-ALL relapse diagnosis
   * Obtention of oral and written consent of the parents
   * Parents affiliated with the social security system
2. Inclusion Criteria for control Group :

   * Children aged from 1 to 18 years enrolled into FRALLE or EORTC treatment protocols, treated for B-ALL and who are in complete molecular remission
   * Obtention of oral and written consent of the parents
   * Parents affiliated with the social security system
3. Exclusion criteria for control Group are the same as for relapsed Group :

   * Children with hematologic syndrome predisposing to hematologic neoplasia (such as Fanconi's anaemia, Diamond Blackfan anaemia …) or acute leukemia secondary to previous treatment, or who have had allogenic hematopoietic stem cell transplantation before relapse

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Measure of Treg (CD4+,CD25+, Foxp3+) and deficient natural killer (NK) cells (CD3-,CD56+,NKp30-) proportions by FACS in children newly diagnosed with their first relapse of B-ALL. | At the time of the inclusion.
  Comparison of the immune status of patients at the diagnosis of their first relapse diagnosis with those of children treated for B-ALL who are in complete remission and at the same stage of treatment.

SECONDARY OUTCOMES:
Measure of the number of T CD4+ lymphocytes (Cluster of Differentiation 4), T CD8+ lymphocytes (Cluster of Differentiation 8), NK cells and Natural killer T (NKT) cells by FACS. | At the time of the inclusion.
Measure of percentage of TCD4+ naive and memory cells and TCD8+ naive and memory cells by FACS. | At the time of the inclusion.
Measure of percentage of gamma delta and alpha-bêta TCR CD3+ T cells by FACS. | At the time of the inclusion.
Measure of TRECs (T cell receptor excision circle) by QPCR and naïve CD4+CD45RA+CD31+ T cells by FACS. | At the time of the inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle PELLIER, PU-PH, Principal Investigator — UNIVERSITY HOSPITAL OF ANGERS
Locations (18):
- France (18):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - University Hospital of Besancon, Besançon
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Caen, Caen
  - Civil Hospices of Lyon, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - University Hospital of Trousseau (Paris), Paris
  - University Hospital of Robert Debre (Paris), Paris
  - University Hospital of Reims, Reims
  - University Hospital of Rennes, Rennes
  - University Hospital of Saint Etienne, Saint-Etienne
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital of Toulouse, Toulouse
  - University Hospital of Tours, Tours